CLINICAL TRIAL: NCT05711030
Title: Thoracic Paravertebral Block Anesthesia for Breast Cancer Surgery: Single-Injection Versus Multiple Injections. A Randomized Controlled Trial
Brief Title: Thoracic Paravertebral Block Anesthesia for Breast Cancer Surgery
Acronym: TPVB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Ariane Clairoux, MD, Principal Investigator, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-3181
Record Dates: First submitted 2022-10-03; First posted 2023-02-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Breast Neoplasms; Breast Neoplasm Female; Cancer, Breast; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Injections

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Blocks will be performed by a different anesthesiologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thoracic paravertebral block multiple (3) injections (Active Comparator): Patients will either be in the sitting or prone position for the block. The block will be performed with the ultrasound transducer in the sagittal position about 2.5 to 3 centimeters (cm) lateral to the spinous process using a caudal to cranial in-plane needle approach. The thoracic vertebral levels will be identified by finding the first rib under ultrasound guidance and counting down levels appropriately.
  The needle (80 mm 22-gauge echogenic SonoPlex needle from Pajunk) will be introduced in-plane in a caudal to cranial direction until it punctures the costotransverse ligament. Saline in 1 ml increments will be injected to confirm correct placement of the needle tip. Injection of saline or local anesthetics deep to the costotransverse ligament will lead to an anterior displacement of the parietal pleura.
  For the 3-level technique, injections will be done at the levels of T2-T3, T3-T4, and T4-T5 with 10 ml of ropivacaine 0.5% at each level.
  Interventions: Procedure: Thoracic paravertebral block multiple (3) injections
- Thoracic paravertebral block single injection (Experimental): Patients will either be in the sitting or prone position for the block. The block will be performed with the ultrasound transducer in the sagittal position about 2.5 to 3 cm lateral to the spinous process using a caudal to cranial in-plane needle approach. The thoracic vertebral levels will be identified by finding the first rib under ultrasound guidance and counting down levels appropriately.
  The needle (80 mm 22-gauge Pajunk) will be introduced in-plane in a caudal to cranial direction until it punctures the costotransverse ligament. Saline in 1 ml increments will be injected to confirm correct placement of the needle tip. Injection of saline or local anesthetics deep to the costotransverse ligament will lead to an anterior displacement of the parietal pleura.
  For the single-injection technique, injection of 30 ml of ropivacaine 0.5% will be done at the T3-T4 paravertebral space after negative aspiration.
  Interventions: Procedure: Thoracic paravertebral block single injection

INTERVENTIONS:
Procedure: Thoracic paravertebral block multiple (3) injections — already described in arm description
  Arms: Thoracic paravertebral block multiple (3) injections
Procedure: Thoracic paravertebral block single injection — already described in arm description
  Arms: Thoracic paravertebral block single injection

SUMMARY:
Background:

Mastectomies are traditionally performed under general anesthesia (GA), often with the addition of regional anesthesia for post-operative pain relief. Thoracic paravertebral blocks (TPVB) had previously been described in the literature to be sufficient for intra-operative anesthesia as an alternative to GA. A 2021 literature review by Cochrane Library comparing paravertebral anesthesia (with or without sedation) to general anesthesia for patients undergoing oncologic breast surgery showed that TPVB could reduce post-operative nausea and vomiting (PONV), hospital stay, postoperative pain and time to ambulation. It also resulted in greater patient satisfaction compared to GA.

The aim of this study is to demonstrate the efficacy of single-injection TPVB done under ultrasound guidance for patients undergoing breast cancer surgery without axillary node dissection.

Hypothesis: Single-injection thoracic paravertebral block is non-inferior to multiple (3) injections for oncologic unilateral breast surgery anesthesia.

Methods: The current study is a prospective randomized controlled trial of patients undergoing oncologic breast surgery without axillary node dissection or immediate reconstruction. Patients will be randomized into two groups; thoracic paravertebral block (TPVB) single-injection or TPVB multiple (three) injections.

Significance/Importance: Oncologic breast surgery performed under TPVB and sedation lowers the risks of post-operative nausea and vomiting, decreases peri-operative use of narcotics, decreases pain scores at rest and on mobilization and leads to better overall patient satisfaction when compared to GA. It also leads to shorter hospital stays. Most studies use multiple injections to perform the block. Even though the risks associated with TPVB are low (3.6 per 1000 surgeries), the single-injection technique could reduce the risks even more. One injection is also easier to perform and of shorter duration, leading to greater patient tolerance and less side effects related to blocks performance duration such as vaso-vagal reactions or general discomfort. To date, no studies have compared the efficacy of single-injection paravertebral block and multiple injection techniques as the main modality of anesthesia for breast cancer surgery.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer among women representing around 25% of new cancer cases worldwide. Surgery is the mainstay of treatment. Mastectomies are usually performed under general anesthesia (GA), often with the addition of regional anesthesia for post-operative pain relief. TPVB have previously been described in the literature to be sufficient for intra-operative anesthesia as an alternative to GA. This technique was first developed by Sellheim in 1905, and was popularized by Eason and Wyatt in 1978. In recent years, there has been a regain of interest for this technique with the easier access to high-performance ultrasound. The thoracic paravertebral space is a wedged shaped space adjacent to the spine bilaterally. It is a continuous space filled with adipose tissue that communicates cranially and caudally. TPVB produce unilateral, segmental, sympathetic and somatic blockade of the chest. Landmark-based techniques were first described, but in recent years ultrasound-guided techniques have been shown to improve the success rate of the block. They can be performed through multiple injections at different thoracic levels or with a single injection. Mutiple injections offer many advantages including coverage for each dermatome associated to the blocked level. Whereas blockade of multiple contiguous levels when performing a single injection implies relying on the spread of local anesthetic (LA) to caudal and cranial levels to block more dermatomes. Some studies have demonstrated that single-injection paravertebral blocks at the level of T3-T4 could be a suitable alternative to general anesthesia, but the blocks were not done under ultrasound guidance and they did not compare the single-injection technique to the multiple injection technique. Thus, a randomized controlled trial comparing the single-injection TPVB technique to the multiple injection technique done under ultrasound guidance for breast cancer surgery anesthesia is needed. The single-injection technique would allow us to offer the TPVB benefits to our patients while decreasing the time to perform the block, the complication rate and therefore potentially improve patient satisfaction.

Our hypothesis is that the TPVB performed as a single injection is non inferior to multiple (three) injections for unilateral oncologic breast surgery without axillary intervention.

The current study is a prospective randomized controlled trial of patients undergoing oncologic breast surgery without axillary node dissection or immediate reconstruction. Patients will be randomized into two groups; thoracic paravertebral block (TPVB) single-injection or TPVB multiple (three) injections. Sedation and analgesia will be standardized for both groups. The block will be performed preemptively by a blinded anesthesiologist at least 20 minutes before surgical incision. 30 milliliters (ml) of ropivacaine 0.5% will be injected on the operating side (maximum 3 milligrams per kilograms (mg/kg)) either as a single injection or fractionated into three injections at three different paravertebral levels.

Preemptive postoperative analgesia plan:

• Each patient will receive standard preemptive postoperative analgesic medication comprising of oral acetaminophen 1 gram (g) preoperatively

Preemptive postoperative nausea and vomiting prevention plan:

• Each patient will receive standard preemptive postoperative nausea and vomiting prevention medication comprising of dexamethasone 4 mg intravenous (IV) at the beginning of the procedure and ondansetron 4 mg IV at the end of the procedure.

Patients will be offered midazolam 1-2 mg IV as needed (PRN) and fentanyl 25-50 mcg IV PRN before performing the TPVB.

All patients will be monitored using 5-lead electrocardiogram, non-invasive blood pressure, pulse oximetry and end-tidal carbon dioxide monitoring. A NOL index (NOL trademark (™), Medasense Biometrics Ltd, Ramat Gan, Israel) as well as a bispectral index device (BIS, Covidien, USA) to allow anesthesia nociception and depth monitoring respectively.

Procedural sedation will be maintained with propofol using BIS monitoring for a target range of 60-80. All patients will receive oxygen (O2) through nasal cannula with end-tidal carbon dioxide (EtCO2) monitoring.

A NOL index monitor will be used to guide analgesic dosage intra-operatively. A NOL > 25 for 1 minute suggests a high nociceptive response. The anesthesiologist will be allowed to give fentanyl in 25 mcg increments every 3 minutes for a maximum of 2 mcg/kg of adjusted body weight. If the maximum dose of fentanyl has been reached, ketamine 0.25 mg/kg can be given and repeated after 10 minutes. If the patient cannot tolerate the surgical procedure after both doses of ketamine have been given, the anesthesiologist will convert to GA by the method of his/her choice.

The total dose of IV fentanyl and ketamine given intraoperatively will be recorded as primary outcomes. Total dose of IV propofol used for sedation will also be recorded.

For the total duration of the anesthesia, monitoring data will be collected electronically via a computer connected to the monitors as well as on the Drager ventilator system. A logbook will be created to allow standardized data collection regarding the primary and secondary endpoints. Total intraoperative fentanyl and ketamine dosages and total postoperative hydromorphone consumption will be recorded. Postoperative hydromorphone will be given in the post-anesthesia care unit (PACU) if the Visual Analog Score (VAS) is > 4/10. Time to meet discharge criteria (Aldrete score > 9) and the incidence of PONV will also be noted.

ELIGIBILITY:
Inclusion Criteria:

• Patients > 18 years old with American Society of Anaesthesiologists (ASA) status I-III, BMI<35, undergoing partial or total mastectomies without axillary lymph node dissection

Exclusion Criteria:

* < 18 years old
* Body mass index (BMI) > 35
* Body weight under 50 kg
* Obstructive sleep apnea (moderate to severe)
* Unable to communicate with the investigators
* Receiving anticoagulation or experiencing any bleeding disorder
* Known allergy to local anesthetics, fentanyl or hydromorphone
* Active infection at injection sites
* Preexisting neurological deficit or psychiatric illness
* Severe cardiovascular disease
* Liver failure
* Renal failure (estimated glomerular filtration rate <15 mL/ min/1.73 m2)
* Pregnancy
* Arrhythmia (NOL monitoring cannot be used reliably)
* Technical inability to proceed with the blocks
* History of chronic pain with daily opioid use during the 3 months before surgery
* Patient refusal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2022-11-04 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Total perioperative fentanyl (mcg) consumption | Intraoperative, about 30 minutes
  To compare the total perioperative fentanyl (mcg) consumption between both groups, using the NOL index to standardize intra-operative dosage and the BIS to standardize propofol sedation. Fentanyl will be given intraoperatively according to the NOL index and the total dose in micrograms will be recorded
Total perioperative ketamine (mg) consumption | Intraoperative, about 30 minutes
  To compare the total perioperative ketamine (mg) consumption between both groups, using the NOL index to standardize intra-operative dosage and the BIS to standardize propofol sedation. Ketamine might be given intraoperatively according to the NOL index (if fentanyl is not sufficient) and the total dose in milligrams will be recorded.

SECONDARY OUTCOMES:
Total dose of propofol (mg) required for sedation | Intraoperative, about 30 minutes
  Total dose of propofol (mg) given during the surgery for a BIS between 60-80
Adverse events | Intraoperative and postoperative, about 3 hours
  Hypotension, vagal reaction during block, Horner's syndrome, bilateral block, bleeding, pleural tap, pneumothorax
Level of the block using ice test preoperatively | Intraoperative, about 30 minutes
  The anesthesiologist will test for block level before proceeding to surgery 20 minutes after the block
Postoperative pain at rest and on movement (VAS) in PACU and day surgery unit | Postoperative, about 2 hours
  VAS score will be recorded in the PACU or day surgery unit every 15 minutes until discharge
Postoperative total analgesic dose of hydromorphone (mg) | Postoperative, about 2 hours
  Total hydromorphone dose (mg) received by each patient will be recorded in the PACU or day surgery unit until discharge
PONV (Post Operative Nausea and Vomiting) in PACU and day surgery unit | Postoperative, about 2 hours
  PONV score (0-3) (A score of 0 meaning no nausea or vomiting, 1 meaning light nausea not requiring treatment, 2 meaning severe nausea requiring treatment and 3 meaning nausea associated with vomiting) will be recorded every 15 minutes in the PACU for each patient as well of the treatment if one was given until discharge
Readiness for hospital discharge (following regular institution criteria) | Postoperative, about 2 hours
  Time of readiness of hospital discharge (Aldrete score >9) will be recorded as well as the time of departure. If there is a difference between those two times, the reason will be noted
Conversion rate to General Anesthesia (GA) | Intraoperative, about 30 minutes
  Conversion rate to GA will be compared between both groups
Block failure rate requiring General Anesthesia (GA) to commence surgery | Intraoperative, about 30 minutes
  Block failure rate will be compared between both groups

CONTACTS AND LOCATIONS:
Overall Officials: Ariane Clairoux, MD, Principal Investigator — Ciusss de L'Est de l'Île de Montréal
Locations (1):
- CIUSSS de l'Est de l'Île de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No